CLINICAL TRIAL: NCT02141607
Title: Multiscale Approach to Describe the Evolution of Molecular Biomarkers in Acute Heart Failure Induced by Shock
Brief Title: Evolution of Molecular Biomarkers in Acute Heart Failure Induced by Shock
Acronym: Shockomics
Status: Completed | Type: Observational
Sponsor: Shockomics Consortium (Network)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Sponsor
Other Study IDs: FP7#602706; 602706 (Other Grant/Funding Number: FP7-HEALTH-2013-INNOVATION-1)
Record Dates: First submitted 2014-05-08; First posted 2014-05-19 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Acute Heart Failure; Shock
Keywords: shock; heart failure; inflammation; biomarkers; cardiovascular instability; metabolic pathways; proteolysis
MeSH Terms: conditions — Shock; Heart Failure; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Hemorrhagic Shock: Hypovolemic shock characterized by:
  * Hypotension: systolic blood pressure < 90 mm Hg or a drop of > 40 mm Hg from baseline or mean arterial pressure < 70 mm Hg persisting despite adequate fluid resuscitation.
  * Rapid loss of significant amount of blood
  * Lactate levels ≥ 2 mmol/L
- Cardiogenic shock: State of inadequate circulation of blood because of ventricular failure due to acute cardiac conditions, concomitant presence of:
  * Hypotension: systolic blood pressure < 90 mm Hg or a drop of > 40 mm Hg from baseline or mean arterial pressure < 70 mm Hg persisting despite adequate fluid resuscitation.
  * Need for a continuous infusion of inotropic drugs
  * Cardiac Index <2.2 L/min/m2 or use of inotropic drugs (dobutamine/isoprenaline/phosphodiesterase inhibitors or levosimendan)
  * Signs of reduced heart function
  * Cardiac overload or altered left/right ventricular function
- Septic shock: Septic shock is defined as sepsis-induced hypotension, defined as systolic blood pressure < 90 mm Hg or a drop of > 40 mm Hg from baseline or mean arterial pressure < 70 mm Hg persisting despite adequate fluid resuscitation.
  Only community medical acquired sepsis with a sepsis onset within 48 hours from hospital admission (i.e. different from nosocomial infection).
  Lactate levels ≥ 2mmol/L.
- control group: The control group will consist on:
  1. 5 healthy blood donors: serving only for the purposes of obtaining reference values for proteomics analysis
  2. a cohort of 20 patients hospitalized for sepsis OR cardiac syndromes not developing shock: will be recruited from patients admitted to the hospital during the study period. The clinical status of the patients will be assessed during hospitalization to ascertain shock and AHF development. Shock development will be an exclusion criteria.

SUMMARY:
The relationship between shock, ischemia and reperfusion (I/R) injury, hemodynamic instability, systemic inflammatory response syndrome and multiorgan failure has been extensively investigated, but there is no consensus on the trigger mechanisms of tissue injury at the molecular level.

Current therapies are targeted to reduce symptoms of shock and multiorgan damage but they are unable to act at the "beginning of the cascade", because of the lack of a model explaining the molecular basis of shock induced tissue injury and ensuing organ damage.

The present observational study is aimed at identifying the molecular triggers of acute heart failure (HF) induced by shock and to identify inflammatory mediators and markers that are activated in shock, with a particular emphasis on the role of uncontrolled proteolytic activity.

ELIGIBILITY:
Inclusion Criteria:

* For patients in septic shock, Severity: SOFA score > 5
* For patients in cardiogenic shock, Severity: SOFA score > 5
* First blood sample available within 16 hours from admission to the ICU.
* Only community medical acquired septic shock. We include patients with shock symptoms and shock diagnosis occurring within the first 48 hours from hospital admission
* Informed Consent available

Exclusion Criteria:

* Risk of rapidly fatal illness and death within 24 hours
* Patients already enrolled in other interventional studies
* N > 4 units of red blood cells transfused
* Patients treated with plasma or whole blood
* Active hematological malignancy
* Metastatic cancer
* Immunodepression, including transplant patients: HIV+, constitutive immune system deficiency, immunosuppressive therapy, systemic corticosteroids (aerosols allowed)
* Patients with pre-existing end stage renal disease needing renal replacement therapy (RRT). The introduction of continuous veno-venous hemofiltration (CVVH), from the day of admission onward is allowed.
* Cardiac surgery patients
* Cirrhosis Child C

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the patients admitted to ICU
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Progression/occurrence of acute heart failure and changes in omics markers in acute phase of shock | within 48 hr after admission in ICU (acute phase of shock)
  The clinical endpoint will be Acute Heart Failure (AHF), assessed by a pool of measures/estimates of cardiac function and filling pressures, based on cardiac output monitoring, inotropic drugs requirements, left and right ventricles assessment using echocardiography.
  The molecular biomarkers changes will be evaluated by means of proteomics, transcriptomics and metabolomics analysis of blood samples collected at the ICU admission and within 48hr after admission.

SECONDARY OUTCOMES:
Progression/Occurence of Acute Heart Failure and changes in omics markers in survivors | within 7 days after admission in ICU (patient stabilization)
  The clinical endpoints will be:
  1. The Acute Heart Failure (AHF) assessed by a pool of measures/estimates of cardiac function and filling pressures, based on cardiac output monitoring, inotropic drugs requirements, left and right ventricles assessment using echocardiography. AHF will be at evaluated within 7 days after ICU admission.
  2. Mechanical ventilation (MV)-free days or organ support (vasopressor, continuous renal replacement therapy (CRRT), etc.) free-days
  3. Survival to ICU
  4. Prognosis at discharge from the ICU (objective - dead or alive, morbidities - and subjective)
  5. Prognosis at discharge from the hospital (objective - dead or alive, morbidities - and subjective).
  The changes in molecular biomarkers will be evaluated by means of proteomics, transcriptomics and metabolomics analysis of blood samples collected within 7 days after ICU admission

OTHER OUTCOMES:
Long term effects of AHF in survivors assessed by changes in omics markers | at about 100 days from ICU admission and enrollment
  Patients discharged after a shock episode have high morbidity and mortality rates, and evidences indicate that physiological condition is restored only after several months. The blood sample will be collected only in patients in healthy conditions, reporting no re-hospitalization associated to shock sequelae during the follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Baselli, MS, Principal Investigator — Politecnico di Milano
Locations (3):
- Department of Intensive Care, Erasme University Hospital, Brussels, Belgium
- Servei de Medicina Intensiva, Hospital Universitari Mútua Terrassa, Barcelona, Spain
- Intensive Care Division, Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carrara M, Bollen Pinto B, Baselli G, Bendjelid K, Ferrario M. Baroreflex Sensitivity and Blood Pressure Variability can Help in Understanding the Different Response to Therapy During Acute Phase of Septic Shock. Shock. 2018 Jul;50(1):78-86. doi: 10.1097/SHK.0000000000001046. PMID 29112634
- [Result] Cambiaghi A, Pinto BB, Brunelli L, Falcetta F, Aletti F, Bendjelid K, Pastorelli R, Ferrario M. Characterization of a metabolomic profile associated with responsiveness to therapy in the acute phase of septic shock. Sci Rep. 2017 Aug 29;7(1):9748. doi: 10.1038/s41598-017-09619-x. PMID 28851978
- [Derived] Maegele M, Aletti F, Efron PA, Relja B, Orfanos SE. NEW INSIGHTS INTO THE PATHOPHYSIOLOGY OF TRAUMA AND HEMORRHAGE. Shock. 2023 Mar 1;59(3S Suppl 1):6-9. doi: 10.1097/SHK.0000000000001954. Epub 2022 Jul 24. PMID 36867756
- [Derived] Braga D, Barcella M, Herpain A, Aletti F, Kistler EB, Bollen Pinto B, Bendjelid K, Barlassina C. A longitudinal study highlights shared aspects of the transcriptomic response to cardiogenic and septic shock. Crit Care. 2019 Dec 19;23(1):414. doi: 10.1186/s13054-019-2670-8. PMID 31856860
- [Derived] Bauza-Martinez J, Aletti F, Pinto BB, Ribas V, Odena MA, Diaz R, Romay E, Ferrer R, Kistler EB, Tedeschi G, Schmid-Schonbein GW, Herpain A, Bendjelid K, de Oliveira E. Proteolysis in septic shock patients: plasma peptidomic patterns are associated with mortality. Br J Anaesth. 2018 Nov;121(5):1065-1074. doi: 10.1016/j.bja.2018.05.072. Epub 2018 Jul 26. PMID 30336851
- [Derived] Aletti F, Conti C, Ferrario M, Ribas V, Bollen Pinto B, Herpain A, Post E, Romay Medina E, Barlassina C, de Oliveira E, Pastorelli R, Tedeschi G, Ristagno G, Taccone FS, Schmid-Schonbein GW, Ferrer R, De Backer D, Bendjelid K, Baselli G. ShockOmics: multiscale approach to the identification of molecular biomarkers in acute heart failure induced by shock. Scand J Trauma Resusc Emerg Med. 2016 Jan 28;24:9. doi: 10.1186/s13049-016-0197-4. PMID 26822963
- [Derived] Carrara M, Baselli G, Ferrario M. Mortality prediction in septic shock patients: Towards new personalized models in critical care. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:2792-5. doi: 10.1109/EMBC.2015.7318971. PMID 26736871